CLINICAL TRIAL: NCT01656954
Title: Change in Stroke Volume During Passive Leg Raise Predicts Volume Challenge Response as Measured by Arterial Pressure Cardiac Output Monitor.
Brief Title: Predicting Volume Response Study
Acronym: PVRS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 813558
Record Dates: First submitted 2012-07-17; First posted 2012-08-03 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2012-07

CONDITIONS: Shock; Hypovolemia
Keywords: stroke volume; cardiac output; pulse pressure variance; stroke volume variance; passive leg raise; fluid challenge; central venous pressure
MeSH Terms: conditions — Shock; Hypovolemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anticipated volume/blood administration: Patients who may receive IV fluid boluses or blood products for restoration of vascular volume. Prior to receiving IV fluid boluses or blood products, the patient will undergo a passive leg raise. (PLR)
  Interventions: Procedure: Passive Leg Raise (PLR)

INTERVENTIONS:
Procedure: Passive Leg Raise (PLR) — From the supine position, the legs are elevated to 45 degrees above the resting surface for a period of 3 minutes. At completion,the legs are lowered to the resting surface.

SUMMARY:
The purpose of this study is to understand and document measurements in heart stroke volume (the volume or amount of blood pumped per heart beat) and cardiac output (the volume or amount of blood pumped by your heart per minute) during a passive leg raise maneuver (elevation of the legs), and to determine if these measurements can predict changes in the same as a result of fluid or blood product administration.

DETAILED DESCRIPTION:
The administration of intravenous fluid and blood products for treatment of hypovolemia is common in the ICU setting. Static resuscitation endpoints such as heart rate, blood pressure, and CVP are frequently used to guide this therapy, despite compelling evidence they are unreliable in predicting patient response to therapeutic volume administration or as an endpoint for ongoing therapy. Dynamic parameters such as continuous stroke volume and cardiac output (index) monitoring, along with pulse pressure and stroke volume variance measures are more reliable in predicting and measuring response to fluid challenge and therapeutic volume administration. The purpose of this study is to observe changes in stroke volume (SV) and cardiac output (CO) during a passive leg raise maneuver (PLR) as a surrogate to volume challenge, and to determine if these changes can predict changes in the same parameters with fluid or blood product administration in surgical patients. The PLR maneuver involves positioning the patient to the supine position and elevating the legs to 45 degrees. The PLR moves blood from the capacitance vessels of the legs to the heart, potentially improving stroke volume (SV) and cardiac output (CO), without the administration of intravenous fluids. PLR may predict whether SV or CO would improve with administration of fluids, and guide decisions on whether fluid administration would be beneficial. Stroke volume and cardiac output (index) will be calculated by a commercial pulse power arterial pressure cardiac output system (LIDCORapid), using the patients' measured heart rate and blood pressure imported from the bedside monitor. By using the combination of a reversible volume challenge (PLR) and a minimally invasive monitoring system, it is hoped that a more reliable method will emerge to both predict a response and guide therapeutic volume administration, while reducing the risk associated with fluid volume overload.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older admitted to the Surgical Intensive Care Unit, anticipated to receive IV fluid boluses or blood products, with the presence of an arterial pressure line.

Exclusion Criteria:

* patients under 18 years of age,
* pregnancy,
* prisoners,
* inability to lay in the supine position,
* conditions of the lower extremities,
* pelvis or spine that preclude elevation of the legs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Rhoads 5 SICU on the Trauma/Surgical Critical Service who would be anticipated to receive IV fluids or blood as part of their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in baseline cardiac stroke volume | Passive Leg Raise: Baseline and at 3 minutes. Fluid/blood administration: Baseline to completion of administration.
  Stroke volume is measured prior to passive leg raise (PLR)and at 3 minutes after completion of the PLR. Stroke volume is measured at baseline after initiation of fluid/blood administration, every 1 minute for 10 minutes, then every 10 minutes until completion of the administration.

SECONDARY OUTCOMES:
Change in baseline stroke volume variance (SVV) | Passive Leg Raise: Baseline and at 3 minutes. Fluid/blood administration: Baseline to completion of administration.
  Stroke volume variance is measured prior to passive leg raise (PLR)and at 3 minutes after completion of the PLR. Stroke volume variance is measured at baseline after initiation of fluid/blood administration, every 1 minute for 10 minutes, then every 10 minutes until completion of the administration.
Change in baseline pulse pressure variance (PPV) | Passive Leg Raise: Baseline and at 3 minutes. Fluid/blood administration: Baseline to completion of administration.
  Pulse pressure variance is measured prior to passive leg raise (PLR)and at 3 minutes after completion of the PLR. Pulse pressure variance is measured at baseline after initiation of fluid/blood administration, every 1 minute for 10 minutes, then every 10 minutes until completion of the administration.
Change in baseline cardiac output | Passive Leg Raise: Baseline and at 3 minutes. Fluid/blood administration: Baseline to completion of administration.
  Cardiac output is measured prior to passive leg raise (PLR)and at 3 minutes after completion of the PLR. Cardiac output is measured at baseline after initiation of fluid/blood administration, every 1 minute for 10 minutes, then every 10 minutes until completion of the administration.
Change from baseline heart rate. | Passive Leg Raise: Baseline and at 3 minutes. Fluid/blood administration: Baseline to completion of administration.
  Heart rate is measured prior to passive leg raise (PLR)and at 3 minutes after completion of the PLR. Heart rate is measured at baseline after initiation of fluid/blood administration, every 1 minute for 10 minutes, then every 10 minutes until completion of the administration.
Change in baseline blood pressure (BP) | Passive Leg Raise: Baseline and at 3 minutes. Fluid/blood administration: Baseline to completion of administration.
  Blood pressure is measured prior to passive leg raise (PLR)and at 3 minutes after completion of the PLR. Blood pressure is measured at baseline after initiation of fluid/blood administration, every 1 minute for 10 minutes, then every 10 minutes until completion of the administration.
Change in baseline central venous pressure (CVP). | Passive Leg Raise: Baseline and at 3 minutes. Fluid/blood administration: Baseline to completion of administration.
  Central venous pressure is measured prior to passive leg raise (PLR)and at 3 minutes after completion of the PLR. Central venous pressure is measured at baseline after initiation of fluid/blood administration, every 1 minute for 10 minutes, then every 10 minutes until completion of the administration.

CONTACTS AND LOCATIONS:
Overall Officials: John J Gallagher, MSN, RN, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States